CLINICAL TRIAL: NCT04845035
Title: A Phase II Study Using a BFM Regimen Plus Tyrosine Kinase Inhibitor in Adult Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: Pediatric-Inspired Chemotherapy Plus Tyrosine Kinase Inhibitor in Adult Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI plans to revise the study design in a new protocol
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.144; HUM00171952 (Other: University of Michigan)
Record Dates: First submitted 2021-04-05; First posted 2021-04-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Dasatinib; Philadelphia chromosome; Ponatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Dasatinib; ponatinib; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BFM + Tyrosine Kinase Inhibitor (Experimental): This study has 2 cohorts: participants aged 18 - 59 years and participants aged 60 or more years. Both cohorts receive the same study intervention with dosage adjusted for age. Participants receive the Berlin-Frankfurt-Münster (BFM) protocol plus dasatinib during a two-phase induction and a delayed re-induction. Participants receive the BFM protocol plus ponatinib during post-induction consolidations and maintenance.
  Interventions: Drug: Dasatinib; Drug: Ponatinib; Drug: Berlin-Frankfurt-Münster Chemotherapy; Drug: Methotrexate and Cytarabine

INTERVENTIONS:
Drug: Dasatinib — By mouth
Drug: Ponatinib — By mouth
Drug: Berlin-Frankfurt-Münster Chemotherapy — with varied cycles, including Daunorubicin, Vincristine, Prednisone, Pegaspargase, Rituximab, Cytarabine, Mercaptopurine, Cyclophosphamide, Methotrexate, Doxorubicin, Thioguanine, and Dexamethasone
Drug: Methotrexate and Cytarabine — Intrathecal

SUMMARY:
This study will combine a standard, pediatric-inspired, chemotherapy regimen with the tyrosine kinase inhibitors (TKIs) Dasatinib and Ponatinib to treat adults with Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia.

There are two age groups/cohorts:

* participants aged 18 to 59 years
* participants aged 60 years and older

One tyrosine kinase inhibitor (TKI), either Dasatinib or Ponatinib, will be administered in each of the respective chemotherapy cycles. The TKI (either Dasatinib or Ponatinib) administered in a given cycle of chemotherapy will be dictated by the given cycle's standard chemotherapy, in order to minimize overlapping side effects of the chemotherapy and TKI.

The dosages of the standard chemotherapy agents, as well as the tyrosine kinase inhibitors (TKIs)--Dasatinib and Ponatinib--have been adjusted for each age group to allow continuous administration of these TKIs.

ELIGIBILITY:
Key Inclusion Criteria

* Patients ≥ 18 years of age.
* Baseline ECOG Performance Status ≤ 2, and patient is a candidate for intensive chemotherapy.
* Newly diagnosed Ph+ ALL.
* Written informed consent prior to any screening procedures. Permitted exceptions are that the diagnostic marrow exam/peripheral blood/nodal biopsy tests confirming Ph+ B-Cell ALL, as well as pre-induction cardiac workup (EKG/TTE/MUGA), may be performed prior to the patient providing written informed consent if these tests are within 14 days of enrollment.
* Patient able to give informed consent.
* B-cell Acute Lymphoblastic Leukemia with BCR-ABL1, i.e., Philadelphia chromosome-positive (Ph+) ALL.

  * B-Cell lineage determined by standard flow cytometry/IHC
  * Ph+ by cytogenetics (karyotype/FISH) and/or molecular (BCR-ABL1 transcripts)
  * Determined in CLIA-certified laboratory
* Previously untreated, except for below allowances in a recent diagnosis and up until 48 hours after starting trial therapy:

  * Corticosteroids
  * Hydroxyurea
  * Leukapheresis

Key Exclusion Criteria

* Any of the following subtypes of ALL:

  * Ph-negative B-Cell ALL.
  * T-Cell ALL.
  * Relapsed Ph+ ALL.
  * Lymphoid blast crisis of chronic myeloid leukemia (CML).
  * Mature B-Cell (Burkitt's) ALL.
* Clinical signs of CNS disease.
* Active ALL in CNS or testes.
* Estimated Glomerular Filtration Rate (eGFR) by MDRD formula and calculated creatinine clearance (CrCl), based on a 24-hour urine collection, < 30 mL/min-unless related to ALL/tumor lysis syndrome and able to be corrected.
* Total Bilirubin > 2x ULN; AST/ALT > 10x ULN, unless related to ALL liver infiltration.
* Patients with known history of HIV, Hepatitis B, or Hepatitis C.
* Pre-treatment QTcF > 480 msecs.
* Left Ventricular Ejection Fraction < 45%. If an initial TTE demonstrates LVEF < 45%, a confirmatory MUGA should be performed to confirm LVEF is < 45% prior to excluding the patient. Both a TTE and a MUGA with LVEF < 45% are needed to exclude a patient. Either a TTE or MUGA alone, if LVEF is ≥ 45%, is sufficient to include a patient.
* Have significant or active cardiovascular disease, specifically including but not restricted to:

  * Known prior type 1 (thrombotic) myocardial infarction (type 2 myocardial infarction/demand ischemia is not necessarily excluded).
  * History of clinically significant atrial arrhythmia or any ventricular arrhythmia.
  * Unstable angina within the last 12 months.
  * Congestive heart failure within the last 12 months.
  * Currently uncontrolled hypertension (≥ Grade 3; or systolic blood pressure ≥ 160 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg).
* Acute pancreatitis within the last year or a history of chronic pancreatitis.
* Have malabsorption syndrome or other gastrointestinal illness that could affect the absorption of orally administered chemotherapy.
* Ongoing uncontrolled severe nausea or vomiting.
* History of a significant bleeding disorder unrelated to ALL, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
* Taking any medications or herbal supplements that are known to be strong inhibitors or inducers of CYP3A4 within at least 7 days or 5 half-lives (whichever is longer) before the first dose of study chemotherapy on day 1 of Remission Induction Phase I (RIP1).
* Active malignancy requiring treatment, other than ALL, within two years prior to start of treatment, with the exception of basal cell or squamous cell carcinoma of the skin, colon polyp, carcinoma in situ of the cervix, or DCIS or LCIS of the breast.
* Active uncontrolled infection, any other concurrent disease, or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator.
* Pregnant women or women who are breast-feeding
* Men and women of childbearing potential must be willing to practice an effective method of birth control during treatment and up until 30 days following the end of trial therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete molecular remission (CMR) at the end of one cycle of Dasatinib + BFM | Post day 36; up to day 43
  CMR will be assessed by minimal residual disease (MRD)-negative status, using quantitative reverse transcription-polymerase chain reaction (RT-qPCR) analysis from bone marrow aspirates, after 1 cycle of induction therapy with Berlin-Frankfurt-Münster (BFM) protocol and Dasatinib.

SECONDARY OUTCOMES:
Rate of Adverse Events related to Dasatinib and Ponatinib | 30 days after last treatment, up to approximately 3 years
  Per NCI CTCAE v5.0 toxicity data, specifically:
  * for dasatinib: pulmonary hypertension (any grade) or grade ≥ 3 serositis/volume overload.
  * for ponatinib: arterial embolism (any grade) and grade ≥ 3 venous thromboembolism, heart failure, or pancreatitis
Percentage of participants who begin ponatinib post-induction that complete at least one cycle. | At 18 weeks
  Feasibility will be assessed by the percentage, among patients who begin the ponatinib post-induction regimen, that complete at least one cycle. Completion is defined as the ability to tolerate ≥ 80% dose intensity of all prescribed anti-cancer agents per cycle of ponatinib initiated.
Complete hematologic (morphologic) remission (CHR) rate after induction | After Remission Induction Phase I and at end of study treatment, up to approximately 3 years
  Bone marrow assessed by morphologic review of both the aspirate smear and core biopsy
Complete cytogenic remission (CCyR) rate post induction | After Remission Induction Phase I and at end of study treatment, up to approximately 3 years
  Bone marrow aspirate assessed by karyotype and/or fluorescence in situ hybridization (FISH).
Complete molecular remission (CMR) rate | After Remission Induction Phase I and at end of study treatment, up to approximately 3 years
  Bone marrow aspirate analyzed by RT-qPCR.
Disease-free survival (DFS) | up to five years after end of study treatment (approximately 8 years)
  Disease-Free Survival (DFS) is defined as the duration of time from attainment of CR (morphologic remission, hematologic remission, etc) to Morphologic Relapse (Relapsed Disease) or Death.
Overall survival (OS). | up to five years after end of study treatment (approximately 8 years)
  Overall Survival (OS) is defined as the length of time from the date of diagnosis that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Burke, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No